CLINICAL TRIAL: NCT01083238
Title: A Phase I, Two-part Study to Investigate the Effects of Food on the PK, Safety and Tolerability of a Single Oral Dose of AZD5069 (120 mg) in Healthy Adult Volunteers (Part A) and to Compare the PK of AZD5069 in Adult and Elderly Healthy Volunteers (Part B)
Brief Title: This Study Will Investigate How Food and Age Effect the Way the Body Handles the AZD5069 Drug Given as a Oral Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D3550C00010
Record Dates: First submitted 2010-02-22; First posted 2010-03-09 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: pharmacokinetics; fasting or after a high fat meal; adult; elderly adult; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Fasting | interventions — N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD5069 following a 10-hour fast
  Interventions: Drug: AZD5069
- 2 (Experimental): AZD5069 30 minutes after the start of a high fat meal
  Interventions: Drug: AZD5069

INTERVENTIONS:
Drug: AZD5069 — 120mg single oral dose

SUMMARY:
AZD5069 is a new drug being tested for the possible treatment of people with chronic obstructive pulmonary disease (COPD).

This is not the first time that AZD5069 will be administered to humans in clinical trials. We are conducting this study to determine whether AZD5069 is safe and well tolerated by healthy males and females in fed and fasted states. We will compare the way the body handles this drug in the fed and fasted states, in subjects in the age group of 18 to 65 years. We will compare the way the body handles this drug between the age groups of 18 to 65 years and above 65 years. We will also be studying how quickly AZD5069 is absorbed into and cleared by the body.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg.

Exclusion Criteria:

* Has participated in another clinical study and received drug treatment within 3 months of the first administration of drug in this study.
* Subjects with a past medical history of tuberculosis (TB).
* Subjects with latent or chronic infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic blood to measure Maximum plasma concentration (Cmax); time to Cmax (tmax); and the area under the plasma concentration-time curve from zero to infinity (AUC). | 0 - 72 hours postdose

SECONDARY OUTCOMES:
Safety and tolerability of AZD5069 by assessing Adverse events, vital signs, electrocardiograms (ECGs), laboratory variables (including high sensitivity C-reactive protein [hsCRP] and circulating neutrophils), blood pressure, pulse rate, body temperature | various timepoints throughout the study from predose to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MBBS DCPSA, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Cullberg M, Arfvidsson C, Larsson B, Malmgren A, Mitchell P, Wahlby Hamren U, Wray H. Pharmacokinetics of the Oral Selective CXCR2 Antagonist AZD5069: A Summary of Eight Phase I Studies in Healthy Volunteers. Drugs R D. 2018 Jun;18(2):149-159. doi: 10.1007/s40268-018-0236-x. PMID 29856004
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1338&filename=D3550C00010_Study_Synopsis.pdf